CLINICAL TRIAL: NCT00612898
Title: A Phase 2b/3, Randomized, Double Blind, Dose Confirming Study of the Safety, Efficacy and Tolerability of Apricitabine Versus Lamivudine in Treatment-experienced HIV-1 Infected Patients With the M184V/I Mutation in Reverse Transcriptase
Brief Title: Study of the Efficacy and Safety of Apricitabine, a New NRTI, to Treat Drug-resistant HIV Infection
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Avexa (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVX-301
Record Dates: First submitted 2008-01-30; First posted 2008-02-12 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: HIV Infections
Keywords: HIV infection; Drug resistance; Reverse transcriptase inhibitor; Nucleoside analogue; treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — apricitabine; Lamivudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 800mg BID apricitabine plus optimised background
  Interventions: Drug: apricitabine
- 2 (Active Comparator): 150mg BID lamivudine plus optimised background
  Interventions: Drug: lamivudine

INTERVENTIONS:
Drug: apricitabine — 800mg BID apricitabine orally for 48 weeks
  Other Names: AVX754
  Arms: 1
Drug: lamivudine — 150mg BID lamivudine orally for 48 weeks
  Other Names: 3TC
  Arms: 2

SUMMARY:
Apricitabine is a new NRTI which is active against drug-resistant HIV. NRTIs are often included as part of patients' treatment, but many HIV-infected patients develop resistance to commonly used NRTIs such as lamivudine (3TC) and emtricitabine (FTC). This study will examine whether including apricitabine as part of patients' treatment is more effective than including lamivudine,when patients change treatment because of drug resistance.

DETAILED DESCRIPTION:
ATC has potent antiviral activity both in vitro (against wild-type HIV-1 and HIV-1 with mutations in reverse transcriptase that confer resistance to NRTIs), and in clinical studies in both treatment-naïve and treatment-experienced patients with M184V, including in the presence of additional NRTI mutations in reverse transcriptase.

The M184V mutation is most commonly present amongst patients failing regimens containing either of the two deoxycytidine analogs lamivudine and emtricitabine. Whilst lamivudine therapy is often maintained in patients harboring the M184V mutation in some settings, there are no deoxycytidine analogs currently available that effectively suppress replication of HIV-1 containing the M184V/I mutation, particularly in the presence of other additional NRTI mutations.

The purpose of this study is to extend the efficacy and safety established in study AVX-201 of ATC in patients who are HIV-1 infected and have failed treatment with lamivudine or emtricitabine and have confirmed M184V/I mutation. Patients to be enrolled will be failing their current lamivudine- or emtricitabine-containing regimen and therefore have limited remaining NRTI treatment options. This study will investigate whether it is possible to improve control of HIV-1 viral replication by including ATC within a treatment experienced patient's new optimized background regimen following ART treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive with M184V/I mutation in reverse transcriptase;
* 18 years of age or older;
* Currently taking lamivudine (3TC) or emtricitabine (FTC)

Exclusion Criteria:

* Female patients who are pregnant or breastfeeding;
* Current hepatitis B virus (HBV) infection;
* Current treatment for hepatitis C virus infection;
* Renal function not adequate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2008-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with plasma HIV-1 RNA <50 copies/mL at W24 | week 24

SECONDARY OUTCOMES:
Time to loss of virological response (TLOVR analysis; FDA algorithm) at W12, W24 and W48 (<50 copies/mL) | week 12, 24, and 48
Proportion of patients with plasma HIV-1 RNA <50 copies/mL at W48 | week 48

CONTACTS AND LOCATIONS:
Overall Officials: Susan W Cox, Ph D, Study Director — Avexa Ltd; Michael Saag, MD, Principal Investigator — UAB Center for AIDS Research
Locations (100):
- United States (33):
  - UAB, 845 19th St South, South Beville Biomedical Research Building, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Southwest Center for HIV/AIDS, Phoenix, Arizona
  - Living Hope Clinical Foundation, Inc, Long Beach, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - AIDS Research Alliance, West Hollywood, California
  - Denver Health & Hospital Authority, Denver, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - George Washington University, Washington D.C., District of Columbia
  - Gary Richmond, MD, Fort Lauderdale, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Infectious Disease Research Institute, Inc, Tampa, Florida
  - Treasure Coast Infectious Diseases Consultants, Vero Beach, Florida
  - Aids Research Consortium Of Atlanta Inc., Atlanta, Georgia
  - Atlanta Infectious Disease Group, PC, Atlanta, Georgia
  - University of Hawaii, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - University of Kansas School of Medicine, Wichita, Kansas
  - Fenway Community Health Center, Boston, Massachusetts
  - Community Research Intiative of New England, Boston, Massachusetts
  - I.D. Care, Inc., Hillsborough, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - Summa Health System, Akron, Ohio
  - The Research & Education Institute, Portland, Oregon
  - Central Texas Clinical Research, Austin, Texas
  - Nicholaos C Bellos, MD, PA, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A., Dallas, Texas
  - Tarrant County Infection Disease Associates, Fort Worth, Texas
  - University of Texas Medical Brach, Galveston, Texas
  - Therapeutic Concepts, Houston, Texas
  - Resarch Access Network, Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Swedish Medical Center, Seattle, Washington
- Australia (8):
  - 407 Doctors, Darlinghurst, New South Wales
  - Parramatta Sexual Health Clinic, Parramatta, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Carlton Clinic, Carlton, Victoria
  - Melbourne Sexual Health Centre, Carlton, Victoria
  - The Alfred, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Prahran Market Clinic, South Yarra, Victoria
- Belgium (3):
  - Prins Leopold Institute voor Tropische Geneeskunde, Antwerp
  - Hopitaux IRIS Sud, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
- Canada (5):
  - Ubc Downtown I.D. Clinic, Vancouver, British Columbia
  - Hamilton Health Sciences Corporation, Hamilton, Ontario
  - University Health Network, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
- Germany (13):
  - EPIMED GmbH, Berlin
  - Charite-Universitatsmedizin Berlin, Berlin
  - Ruhr-Universitat Bochum, Bochum
  - Universitatsklinikum Bonn, Bonn
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitatsklinikum Essen, Essen
  - Klinikum der Johann-Wolfgang Goethe-Universitat, Frankfurt
  - Praxis fuer Innere Medizin, Freiburg im Breisgau
  - Praxis Dr.Schneider, Fürth
  - Dr. med. Birger Kuhlmann, Hanover
  - Klinikum der Universitat Munchen - Innenstadt, München
  - Gemeinschaftspraxis E. Schnaitmann, Dr. med. A. Schaffert, Dr. med. A. Trein, Dr. med. E. Ibler, Stuttgart
  - Praxis Dres. Ulmer, Frietsch, Muller, Stuttgart
- Israel (6):
  - Soroka University Medical Center, Beersheba
  - Rambam Medical Center, Haifa
  - Hadassah University Hospital Ein Kerem, Jerusalem
  - The Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - Ospedale S.Maria Annunziata, Antella
  - Azienda Ospedaliera Universitaria di Ferrara Arcispedale S.Anna, Ferrara
  - Azienda Ospedaliera Universitaria San Martino, Genova
  - Fondazione Centro San Raffaele del Monte Tabor, Milan
  - Ospedale Luigi Sacco, Milan
  - Azienda Ospedaliero-Universitaria di Modena Policlinico, Modena
  - Azienda Ospedaliera Cotugno, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Istituto Nazionale Malattie Infettive "Lazzaro Spallanzani" IRCCS, Roma
  - Comprensorio Amedeo di Savoia - Birago Di Vische, Torino
- Peru (6):
  - Hospital Nacional CASE-EsSalud, Arequipa
  - Investigaciones Medicas en Salud, Lima
  - Hospital Dos de Mayo, Lima
  - Via Libre, Lima
  - Hospital Nacional Cayetano Heredia, Lima
  - Edgardo Rebagliati Hospital, Lima
- Puerto Rico (3):
  - Instituto De Investigacion Cientifica, Ponce
  - University of Puerto Rico, San Juan
  - Hope Clinical Research, San Juan
- Thailand (8):
  - Mahidol University Hospital for Tropical Diseases, Bangkok
  - Pharmongkutklao Hospital, Bangkok
  - The HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT), Bangkok
  - Ramathibodi Hospital, Mahidol University, Bangkok
  - Sirraj Hospital, Mahidol Universoty, Bangkok
  - Maharaj Nakorn Chiang Mai, Chiang Mai University, Chiang Mai
  - Khon Kaen University, Khon Kaen
  - Bamrasnaradura Institution, Nonthaburi
- United Kingdom (5):
  - Birmingham Heartlands Hospital, Birmingham
  - St Bartholomew's Hospital, London
  - Royal Free Hospital, London
  - Guy's King's & St. Thomas' School of Medicine, London
  - St Mary's Hospital, London